CLINICAL TRIAL: NCT03994419
Title: PErioperAtive CHildhood obesitY (PEACHY): A Prospective Observational Cohort Study Investigating the Proportion of Overweight and Obese Children Presenting for a Procedure Under General Anaesthesia in the UK and the Incidence of Perioperative Adverse Outcomes in This Patient Group
Brief Title: PErioperAtive CHildhood ObesitY
Acronym: PEACHY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Association of Paediatric Anaesthetists of Great Britain & Ireland (APAGBI) (Unknown); University of Aberdeen (Other); Paediatric Anaesthesia Trainee Research Network (PATRN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS 248493
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Pediatric Obesity; Obesity, Childhood; Overweight and Obesity; Perioperative/Postoperative Complications
Keywords: Paediatric; Anaesthesia
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Postoperative Complications | interventions — Anesthesia; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Anaesthesia for surgery — Observational study observing proportion of obese and overweight children attending for surgery. Observing adverse events following general anaesthesia for surgery in obese versus healthy weight children.

SUMMARY:
The incidence of childhood obesity is at epidemic levels and increasing in the UK. Obese adults are considered a high-risk group of patients for general anaesthesia with published national guidelines on the best practice management. The proportion of children presenting for a procedure under general anaesthesia in the UK who are overweight or obese is currently unknown.

Obese children are perceived to be at greater risk of complications from general anaesthesia. Previous non-UK studies suggest they take longer to recover from anaesthesia, require more medications to combat nausea and vomiting and are at greater risk of complications that may threaten their airway and breathing.

This study involves reviewing the anaesthetic care record and patient notes to collect information relating to general anaesthesia and basic demographic data in children aged 2-16 years presenting for a procedure under general anaesthesia.

The aims of this study are to establish the prevalence of obesity in the paediatric surgical population (i.e. the proportion of children attending UK hospitals for procedures under general anaesthesia who are overweight or obese) and to ascertain whether obese children are at increased risk compared to their healthy weight counterparts.

This information will be used with the goal of reducing avoidable harm both at national and local level in the future.

DETAILED DESCRIPTION:
IRAS 248493 REC 18/WM/0394 NIHR CPMS ID 40368

Hypotheses

1. Overweight and obese children commonly present for procedures under general anaesthesia.
2. Obese children are at higher risk of perioperative adverse events compared to their healthy-weight counterparts.
3. There is wide variation in paracetamol drug dosing amongst obese children.
4. Obese children may be more likely to present for certain surgery compared to their healthy-weight counterparts.

This observational cohort study will take place in NHS hospitals in the UK with trainee anaesthetists affiliated to the Paediatric Anaesthesia Trainee Research Network (PATRN). To increase coverage of sites in the UK, the project will be advertised through other trainee research networks including Research and Audit Federation of Trainees (RAFT) and through the Association of Paediatric Anaesthetists of Great Britain and Ireland (APAGBI) linkmen.

Each hospital taking part will have a nominated anaesthetic consultant and trainees who will act as local investigators collecting data. Data will be collected for all children aged 2-16 years weighing >12kg presenting for a procedure involving general anaesthesia during the defined study period. This will be one week (7 consecutive days). Using previous PATRN audit projects as a guide, we aim to enrol approximately 90 local sites which will give an estimated total of 7590 children attending for a procedure under general anaesthesia during the study period.

Patients will be identified by local trainee investigators (independent of delivery of anaesthesia but part of the anaesthetic department of the hospital) from operating department lists on the days of the study. Data will be collected on all eligible patients who undergo a procedure under general anaesthesia during the study period. Similar data collection tools have been used in previous PATRN audit projects.

Data will be collected from the paper or electronic anaesthetic record and clinical notes. Only routine clinical data will be included and where this is unavailable the domain will be left blank. Data will be collected using a single paper case report form (CRF) per patient. This will be initiated by the anaesthetist in the operating theatre and completed by recovery staff in PACU. Patient identifiable data in the form of hospital number and date of birth will be collected on the CRF for traceability in terms of missing data.

To calculate BMI, age (to the nearest month), gender, height and weight are required for each patient. It is anticipated that all hospitals would routinely measure weight but some hospitals may not routinely measure height prior to a procedure under general anaesthesia. NICE guidelines currently recommend that clinical judgement should be used to decide when to measure a person's height and weight, including at routine health checks. The preoperative setting is a specific health check prior to undergoing general anaesthesia and therefore an appropriate time to measure a child's height and weight.

Height will be measured with shoes removed to the nearest 0.1cm using a height measure with the child's head positioned so that the Frankfurt plane is horizontal. Body weight will be measured with patients lightly clad, to the nearest 0.1kg using a calibrated electronic weighing scale. If the local site is unable to collect age, gender, height and weight we will ask for the case to be logged and uploaded but for no other data to be collected. It is important to know how many cases we are unable to include in the analysis due to incomplete data.

Other information that would routinely be recorded within the clinical notes relating to the patients physical status, surgery, anaesthetic and specific perioperative adverse events will also be collected on the CRF.

The completed CRF will be taken directly to a secure location accessible by the local investigator. The data will be entered electronically via a secure encrypted connection into an online portal managed by Aberdeen University. The software used for data capture will be REDCap (Research Electronic Data Capture - http://www.project-redcap.org). REDCap is a mature, secure web application for building and managing online surveys and databases.

Each dataset entered will generate a unique identifier (ie the data will be pseudonymised); local investigators will be asked to keep a log of their unique identifiers linked to local hospital identification numbers. The hospital number will remain within the respective trusts, meaning only the local NHS staff responsible for care have access to personal identifying information. The study database will be closed for data entry a number of weeks after the study completion date. The anonymised responses from participating hospitals across the country will be analysed by a team of researchers.

ELIGIBILITY:
Inclusion Criteria:

* All children aged greater than or equal to two years and less than 16 years presenting for a procedure under general anaesthesia.
* Elective cases, day case and emergency cases will all be included.
* Private cases being undertaken in NHS hospitals will be included.
* MRI, radiology, oncology and dental cases will be included provided the patient receives a general anaesthetic.

Exclusion Criteria:

* Procedures performed under sedation or local anaesthesia.
* Children aged less than two years since the 0-24 month age group has separate growth charts, which are not currently recommended for interpretation of BMI.
* Children weighing less than 12kg as these are not included on the growth charts for interpretation of BMI.
* Children requiring general anaesthesia purely as part of intensive care treatment.
* Children who are already anaesthetised in the intensive care setting being transferred for a scan or procedure without any intervention to their airway planned.
* Children 16 years or more may be counted as children in some hospitals but not for the purposes of this study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children aged 2-16 years and weighing >12kg presenting for a procedure under general anaesthesia in registered sites across the UK (England, Wales, Scotland and Northern Ireland) during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2019-09-09 (Estimated); Primary Completion 2019-10-06 (Estimated); Study Completion 2019-10-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of overweight and obesity in UK children attending for surgery | One week study period
  The proportion of overweight and obesity in UK children aged 2-16 years attending hospitals for a procedure under general anaesthesia.

SECONDARY OUTCOMES:
Adverse events | One week study period
  The proportion of defined adverse events occurring in obese children as compared to healthy weight children attending for a procedure under general anaesthesia.
Paracetamol dosing variation | One week study period
  The variation in paracetamol dosing in obese children in the UK perioperative setting.
Surgery types | One week study period
  The proportion of obese children presenting for certain types of surgery compared to their healthy weight counterparts.
Comparison with the UK National Child Measurement Programme | One week study period
  The difference in the proportion of overweight and obesity in the perioperative setting compared to that from the UK National Child Measurement Programme (NCMP).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Edwards, Principal Investigator — University Hospital Southampton NHS Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton ZA, Lewis R, Bennett T, McLernon DJ; Paediatric Anaesthesia Trainee Research Network; Engelhardt T, Brooks PB, Edwards MR. Prevalence of PErioperAtive CHildhood obesitY in children undergoing general anaesthesia in the UK: a prospective, multicentre, observational cohort study. Br J Anaesth. 2021 Dec;127(6):953-961. doi: 10.1016/j.bja.2021.07.034. Epub 2021 Oct 6. PMID 34627621